CLINICAL TRIAL: NCT07374783
Title: The Effect of Sensory Isolation on Physiological Indicators of Anxiety in Patients Undergoing Fiberoptic Bronchoscopy: A Randomized Controlled Trial
Brief Title: Sensory Isolation to Reduce Anxiety During Bronchoscopy
Acronym: Bronchoscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Melek YÜKSEL (Other)
Collaborators: Ege University (Other)
Responsible Party: Sponsor-Investigator, Melek YÜKSEL, Ege University Faculty of Nursing, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EGE-BRONCH-2025-01
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Anxiety Physiological Stress Responses ,Fiberoptic Bronchoscopy, Sensory Isolation
Keywords: Sensory isolation Anxiety Physiological responses Nursing intervention Randomized controlled trial, Pre-procedural anxiety, Nonpharmacological intervention
MeSH Terms: interventions — Ear Protective Devices

STUDY DESIGN:
Intervention Model Description: This study follows a parallel-group, randomized controlled design. Participants who meet the inclusion criteria will be assigned in a 1:1 ratio to either the intervention group (sensory isolation using an eye mask and earplugs) or the control group (standard care). Randomization will be stratified by age group (under 65 years and 65 years and older) and gender to ensure balanced group distribution.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - Sensory Isolation (Experimental): Participants in this group will receive sensory isolation using an eye mask and earplugs applied approximately 10 minutes before and during the fiberoptic bronchoscopy procedure. Physiological parameters (blood pressure, heart rate, respiratory rate, and oxygen saturation) and anxiety levels will be assessed at predefined time points before, during, and after the procedure.
  Interventions: Behavioral: Sensory Isolation (Eye Mask and Earplugs)
- Control Group - Standard Care (No Intervention): Participants in this group will receive routine standard care during fiberoptic bronchoscopy without the use of sensory isolation tools. Anxiety levels and physiological parameters will be assessed at the same predefined time points as in the intervention group.

INTERVENTIONS:
Behavioral: Sensory Isolation (Eye Mask and Earplugs) — Participants assigned to the intervention group will receive sensory isolation using an eye mask and earplugs applied approximately 10 minutes before and during the fiberoptic bronchoscopy procedure. This is a non-pharmacological behavioral nursing intervention intended to minimize exposure to visual and auditory stimuli. Anxiety levels and physiological parameters will be assessed at predefined time points before, during, and after the procedure.
  Other Names: Eye mask and earplug intervention; Sensory isolation
  Arms: Intervention Group - Sensory Isolation

SUMMARY:
TThis randomized controlled trial aims to evaluate the effect of sensory isolation on anxiety and physiological parameters in patients undergoing fiberoptic bronchoscopy. The intervention involves the use of an eye mask and earplugs to reduce environmental stimuli. The study will comparatively assess the effects of sensory isolation on anxiety levels and physiological parameters, including blood pressure, heart rate, and oxygen saturation.

DETAILED DESCRIPTION:
This study is designed as a parallel-group, randomized controlled trial to evaluate the effect of sensory isolation on anxiety and physiological parameters in patients undergoing fiberoptic bronchoscopy. The research will be conducted at the Ege University Faculty of Medicine, Department of Chest Diseases, Bronchoscopy Unit, and the Suat Seren Chest Diseases and Thoracic Surgery Training and Research Hospital.

Participants who meet the inclusion criteria and provide written informed consent will be randomly assigned in a 1:1 ratio to either the intervention group (sensory isolation using an eye mask and earplugs) or the control group (standard care). To ensure balanced distribution between groups and to minimize potential confounding effects on anxiety and physiological responses, stratified block randomization will be applied based on age group (under 65 years and 65 years and older) and gender. Within each stratum, randomization sequences will be generated using Random.org (List Randomizer) with a fixed block size of six (3 intervention, 3 control).

Allocation concealment will be ensured through the use of sequentially numbered, opaque, sealed envelopes prepared separately for each stratum. At the time of enrollment, participants will be assigned to groups according to the next envelope in sequence, thereby preventing foreknowledge of group allocation and minimizing selection bias.

The randomization and reporting processes of the study will be conducted in accordance with the CONSORT (Consolidated Standards of Reporting Trials) 2025 guidelines to ensure methodological rigor, internal validity, and transparency.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing fiberoptic bronchoscopy (FOB) for the first time.
* Aged 18 years or older.
* Able to read and understand written study materials.
* Willing to participate and able to provide written informed consent.
* Able to communicate effectively and cooperate during data collection.
* Undergoing fiberoptic bronchoscopy under local anesthesia only, without general anesthesia or procedural sedation.

Exclusion Criteria:

* Patients requiring emergency bronchoscopy.
* Patients requiring endotracheal intubation or invasive mechanical ventilation during the procedure.
* Patients who withdraw consent or are unable to comply with the study protocol.
* Patients with a diagnosed psychiatric disorder that may affect anxiety assessment.
* Patients with dementia or other cognitive impairments affecting comprehension or cooperation.
* Patients with severe cardiovascular disease, including advanced heart failure.
* Individuals with hearing or visual impairments that interfere with the application of sensory isolation procedures.
* Patients whose fiberoptic bronchoscopy procedure exceeds 10 minutes in duration.fiberoptic bronchoscopy lasts longer than 10 minutes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-07-20 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety level (State Anxiety Inventory - STAI) | Baseline (10 minutes before bronchoscopy) and end of procedure (10th minute)
  Anxiety will be assessed using the State Anxiety Inventory (STAI; score range 20-80, with higher scores indicating greater anxiety). Anxiety levels will be compared between the intervention and control groups to evaluate the effect of sensory isolation during fiberoptic bronchoscopy.

SECONDARY OUTCOMES:
Heart rate | 10 minutes before, start of procedure (0 min), 5th minute, end of procedure (10th minute), and 20 minutes after the procedure
  Heart rate will be measured using standard clinical monitoring to assess physiological stress responses during fiberoptic bronchoscopy.
Systolic blood pressure | 10 minutes before, 0 min, 5 min, 10 min, and 20 min post-procedure
  Systolic blood pressure will be measured using automated monitors to evaluate hemodynamic responses during the procedure.
Diastolic blood pressure | 10 minutes before, 0 min, 5 min, 10 min, and 20 min post-procedure
  Diastolic blood pressure will be measured using automated monitors to evaluate hemodynamic responses during the procedure.
Respiratory rate | 10 minutes before, 0 min, 5 min, 10 min, and 20 min post-procedure
  Respiratory rate will be measured to evaluate respiratory stress responses during fiberoptic bronchoscopy.
Oxygen saturation (SpO₂) | 10 minutes before, 0 min, 5 min, 10 min, and 20 min post-procedure
  Peripheral oxygen saturation will be measured using standard pulse oximetry to detect changes during fiberoptic bronchoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla KHORSHİD, PhD, Study Director — Ege University, Faculty of Nursing
Locations (2):
- Turkey (Türkiye) (2):
  - Ege University Faculty of Medicine, Department of Chest Diseases, Bronchoscopy Unit, Izmir
  - Suat Seren Chest Diseases and Thoracic Surgery Training and Research Hospital, Izmir

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves patient-specific clinical and psychological data collected under institutional ethics approval. Data sharing is restricted to protect participant confidentiality in accordance with national and international data protection regulations (KVKK/GDPR). Only aggregated and fully anonymized results will be disseminated through scientific publications and academic presentations.